CLINICAL TRIAL: NCT06758375
Title: Low-dose Teclistamab As Consolidation in the First-line Treatment of Patients with Newly Diagnosed Multiple Myeloma.
Brief Title: Low Dose Teclistamab in Newly Diagnosed Multiple Myeloma Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, David Gomez Almaguer, Chief of the Hematology Service, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE24-00015
Record Dates: First submitted 2024-12-22; First posted 2025-01-03 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma, Newly Diagnosed
Keywords: Multiple myeloma; Teclistamab; Newly diagnosed multiple myeloma; Low-dose teclistamab
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: One arm, open-label, phase 2 study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): Patients receiving 3 cycles of VRd followed by low-dose teclistamab.
  Interventions: Drug: Low-dose teclistamab

INTERVENTIONS:
Drug: Low-dose teclistamab — NDMM patients will receive VRd 3x cicles followed by low dose teclistamab.

SUMMARY:
This single-arm, open-label study aims to determine the efficacy and safety of low-dose, limited-duration teclistamab as a consolidation scheme in newly diagnosed multiple myeloma (NDMM) patients.

DETAILED DESCRIPTION:
This single-arm, open-label study aims to determine the efficacy and safety of low-dose (1.0 mg/kg), limited-duration teclistamab as a consolidation scheme in newly diagnosed multiple myeloma (NDMM) patients after 3 (three) VRd cycles as induction therapy.

Patients with MMND who meet the established inclusion criteria will be invited to participate. A single-arm phase 2 study will be conducted in the Hematology Department of the University Hospital, where an induction schedule of 3 cycles of bortezomib, lenalidomide, and dexamethasone (VRd) will be administered followed by consolidation with 4 therapeutic doses of teclistamab at 1.0 mg/kg subcutaneously. Four weeks after the last dose of teclistamab, the clinical response will be assessed according to standard International Myeloma Working Group (IMWG) criteria. Those with a complete response (CR) or better will be assessed for measurable residual disease (MRD) with multiparametric flow cytometry with a sensitivity of 10^6. Patients with CR and negative MRD will be kept under active surveillance for 18 months, while those with positive MRD or high cytogenetic risk will be offered biweekly bortezomib as maintenance. On the other hand, patients with very good partial response (VGPR) or worse will be offered 1-2 additional therapeutic doses of teclistamab and reevaluated 4 weeks after the last dose. Finally, patients who do not achieve CR will exit the study and will continue their management according to the standard of care recommended by their treating physician.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age.
* Newly diagnosed multiple myeloma.
* Eastern Cooperative Oncology Group (ECOG) Performance Status Score of 0 or 1.
* Women of childbearing potential must have a negative serum pregnancy test prior to starting treatment and agree to use a highly effective method of contraception, such as a hormonal method that inhibits ovulation, an intrauterine device, or a vasectomy partner.
* Males: agree to use a highly effective contraceptive method, such as a male condom or vasectomy.

Exclusion Criteria:

* History of previous treatment for MM.
* Active central nervous system (CNS) involvement or clinical signs of meningeal involvement of multiple myeloma.
* Plasma cell leukemia, Waldenström's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin changes) or AL amyloidosis.
* Severe active infection secondary to viruses, bacteria or fungi.
* Pulmonary disease requiring supplemental oxygen.
* History of allogeneic or autologous hematopoietic cell transplantation.
* Vaccination with live attenuated virus in the 4 weeks prior to teclistamab administration.
* Major surgery during the 2 weeks prior to the first dose or absence of complete recovery from surgery.
* Presence of other concomitant malignancy.
* Hepatitis B and C virus infection or human immunodeficiency virus (HIV) infection.
* Cerebrovascular events or seizures in the last 6 months.
* Congestive heart failure class III-IV according to NYHA (New York Heart Association Stage).
* Acute myocardial infarction or history of coronary revascularization surgery in the last 6 months.
* Women of childbearing age: active pregnancy prior to the first administration of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-09-07 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
To determine general response | 18 months after last teclistamab dose
  Evaluated according to the IMWG response criteria including MRD status.

SECONDARY OUTCOMES:
To determine response duration | Up to 18 months after last teclistamab dose
  Evaluated according to the IMWG response criteria including MRD status.
Adverse events | Through the study completion and up to 18 months after last teclistamab dose
  To report the side effects related to the trial's treatment as per the international guidelines for chemo- and immunotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Dr. Jose E. Gonzalez, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Girgis S, Lin SXW, Pillarisetti K, Banerjee A, Stephenson T, Ma X, Shetty S, Yang TY, Hilder BW, Jiao Q, Hanna B, Adams HC 3rd, Sun YN, Sharma A, Smit J, Infante JR, Goldberg JD, Elsayed Y. Translational Modeling Predicts Efficacious Therapeutic Dosing Range of Teclistamab for Multiple Myeloma. Target Oncol. 2022 Jul;17(4):433-439. doi: 10.1007/s11523-022-00893-y. Epub 2022 Jun 24. PMID 35749004
- [Background] Usmani SZ, Garfall AL, van de Donk NWCJ, Nahi H, San-Miguel JF, Oriol A, Rosinol L, Chari A, Bhutani M, Karlin L, Benboubker L, Pei L, Verona R, Girgis S, Stephenson T, Elsayed Y, Infante J, Goldberg JD, Banerjee A, Mateos MV, Krishnan A. Teclistamab, a B-cell maturation antigen x CD3 bispecific antibody, in patients with relapsed or refractory multiple myeloma (MajesTEC-1): a multicentre, open-label, single-arm, phase 1 study. Lancet. 2021 Aug 21;398(10301):665-674. doi: 10.1016/S0140-6736(21)01338-6. Epub 2021 Aug 10. PMID 34388396